CLINICAL TRIAL: NCT06929702
Title: Early Model-Informed Precision Dosing of Beta-lactam Antibiotics in Critically Ill Children: Big Solution for Small People?
Brief Title: Precision Dosing of Beta-lactam Antibiotics in Critically Ill Children
Acronym: MOMENTUM
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2024-0295; 2024-516447-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-13; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Amoxicillin-clavulanate; Piperacillin-tazobactam; Meropenem
Keywords: amoxicillin-clavulanate; piperacillint-tazobactam; meropenem; model-informed precision dosing; dose calculator; critically ill children
MeSH Terms: interventions — Monobactams; Amoxicillin-Potassium Clavulanate Combination; Piperacillin, Tazobactam Drug Combination; Meropenem

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and legal representatives are blinded for the allocation to the intervention or standard-of-care arm until the end of study. The statistician is kept blinded until after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care beta-lactam treatment (Active Comparator): Beta-lactam standard-of-care dosing regimen, as currently used at participating wards, during 28 day study period
  Interventions: Drug: Beta-lactam antibiotic
- Beta-lactam model-informed precision dosing (Experimental): fT>MIC-based model-informed precision dosing of beta-lactam antibiotics using a dosing calculator during 28 day study period.
  Interventions: Drug: Beta-lactam antibiotic; Device: Beta-lactam model-informed precision dosing

INTERVENTIONS:
Drug: Beta-lactam antibiotic — amoxicillin-clavulanic acid, piperacillin-tazobactam, meropenem treatment
  Other Names: amoxicillin-clavulanic acid; piperacillin-tazobactam; meropenem
Device: Beta-lactam model-informed precision dosing — A dosing calculator is used for the prediction of starting doses (a priori dose predictions) and follow-up doses (a posteriori calculations), using a target 100% fT>MIC.
  Other Names: Dosing calculator
  Arms: Beta-lactam model-informed precision dosing

SUMMARY:
The overall objective of this study is to investigate the impact of early model-informed precision dosing (MIPD) on target attainment of three beta-lactam antibiotics (amoxicillin-clavulanic acid, piperacillin-tazobactam and meropenem) in critically ill children. This evaluation includes a comparison with the more standard approach on clinical and patient-oriented measures.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged between 0 - 17 years 10 months.
* Subject admitted to a participating ward unit (Neonatal Intensive Care Unit, Pediatric Intensive Care Unit, Pediatric Hematology-Oncology unit).
* Strongly suspected or confirmed systemic infection.
* Subject planned to start on intravenous amoxicillin-clavulanic acid, piperacillin-tazobactam or meropenem treatment at least aimed for a minimum duration of two days at time of inclusion. If the subject was previously treated with the same beta-lactam, the minimum interval to the previous beta-lactam treatment episode is
* 40 hours for amoxicillin-clavulanic acid (based on elimination half-life)
* 8 hours for piperacillin-tazobactam and meropenem (based on elimination half-life) Subject planned to start on intravenous amoxicillin (without clavulanic acid) will not be included.
* Informed consent/assent signed by parents or legal representatives of the subject.
* Not previously enrolled in this trial.

Exclusion Criteria:

* Subject with serum creatinine level ≥ 2 mg/L at inclusion.
* Subject receiving (or planned to receive) haemofiltration, extracorporeal membrane oxygenation, hemodialysis or peritoneal dialysis, molecular adsorbent recirculating system or any other exchange technique.
* Subject receiving (or planned to receive) body cooling.
* Subject death is deemed imminent and inevitable.
* Reporting of first dosing advice (based on blood sampling) is not possible within 28 hours (*) after start treatment.
* The subject is known or suspected to be pregnant.
* The subject has a known allergy to the specific beta-lactam antibiotic.

(*) The first (a posteriori) dose calculation and dose adjustment if necessary, is performed within a maximum timeframe of 28 hours after start of treatment (i.e. maximum timeframe to first dose adjustment).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-22 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects reaching the therapeutic target 100% fT>MIC | At 48 hours after start of beta-lactam treatment
  fT>MIC refers to the percentage of the dosing interval during which the beta-lactam concentration remains above the Minimum Inhibitory Concentration (MIC).
  A target lower boundary for trough concentrations is set to achieve 100% fT>MIC.
  A conservative upper threshold for trough concentrations of 100% fT>4xMIC is used.
  Therefore, the therapeutic target range is 10-40 mg/L for amoxicillin (*), 18-72 mg/L for piperacillin (**) and 2-8 mg/L for meropenem (***).
  (*) 10 mg/L for amoxicillin: taking into account a EUCAST breakpoint (for Escherichia coli infections) of 8 mg/L and a plasma protein binding of 18%.
  (**) 18 mg/L for piperacillin: taking into account a EUCAST breakpoint (for wild-type Pseudomonas spp. infections) of 16 mg/L and a plasma protein binding of 9%.
  (***) 2 mg/L for meropenem: taking into account a EUCAST breakpoint of 2 mg/L (for wild-type Enterobacterales species) and a plasma protein binding of 2%.

SECONDARY OUTCOMES:
Proportion of subjects reaching the therapeutic target 100% fT>MIC | At 120 hours after start of beta-lactam treatment
  The therapeutic target range is 10-40 mg/L for amoxicillin, 18-72 mg/L for piperacillin and 2-8 mg/L for meropenem.
Proportion of subjects reaching the therapeutic target 100% fT>MIC | Within the interval 48 to 72 hours after start of beta-treatment
  The therapeutic target range is 10-40 mg/L for amoxicillin, 18-72 mg/L for piperacillin and 2-8 mg/L for meropenem.
Hospital length-of-stay | From date of randomization until date of hospital discharge, with a maximum of 28 days.
  Number of days from randomization to hospital discharge. Patients who are not discharged from hospital within 28 days will be censored at 28 days, the maximum follow up time. Patients who die before hospital discharge will also be censored at 28 days.

OTHER OUTCOMES:
Proportion of subjects with supratherapeutic beta-lactam concentration | At 48 hours and at 120 hours after start of beta-lactam treatment
  A supratherapeutic concentration is defined as > 40 mg/L for amoxicillin, > 72 mg/L for piperacillin and > 8 mg/L for meropenem.
Mean percentage of time above the therapeutic target 100% fT>MIC | Within the interval 0 hours (baseline) to 120 hours (Day 5) after start of beta-treatment.
  Above the therapeutic target is defined as > 10 mg/L for amoxicillin, > 18 mg/L for piperacillin and > 2 mg/L for meropenem.
Proportion of subjects with clinical cure | At day 14 after start of beta-lactam treatment
  Clinical cure will be defined as the completion of the beta-lactam treatment course (on or prior to test-of-cure day 14) without recommencement of antibiotic therapy within 48 hours of cessation. Change of antibiotic therapy (i.e. either escalation or de-escalation) for the same indication for which the beta-lactam antibiotic was commenced is considered part of the antibiotic treatment course. Participants discharged from the hospital within 14 days after start of beta-lactam antibiotic will be considered to meet the definition of clinical cure.
Number and type of adverse events and serious adverse events, considered to be related to study assigned dosing method (possibly, probably or definitely) | From start date of beta-lactam treatment until stop date of beta-lactam treatment (up to 28 days)
Feasibility and compliance endpoint: time elapsed from blood collection to TDM concentration result availability | Blood samples taken within 120 hours of starting beta-lactam treatment (0-120 hours)
  Blood samples will be collected within the first five days (120 hours) after starting beta-lactam treatment. A maximum of 8 blood samples will be taken from subjects in both the control and intervention group.
Feasibility and compliance endpoint: time elapsed from first dose of antimicrobial to TDM concentration result availability | The first two blood samples are collected within a maximum timeframe of 24 hours after start of beta-lactam treatment. TDM concentration is measured once a day and only on weekdays.
Feasibility and compliance endpoint: number of possible dose adjustments | At 48 hours after start of beta-lactam treatment
  Number of times a dose could be adjusted based on the TDM concentration result. Three blood samples are taken within 48 hours after start of beta-lactam treatment: The first two blood samples are collected within a maximum timeframe of 24 hours after start of treatment. One random sample is taken between 24 and 48 hours after start of treatment.
Feasibility and compliance endpoint: Proportion of dosing advices implemented (before the next planned dose) by the prescriber | From start date of beta-lactam treatment until stop date of beta-lactam treatment (up to 28 days).

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Dhont, Dr., Principal Investigator — Ghent University Hospital, Princess Elisabeth Children's Hospital
Locations (1):
- Ghent University Hospital, Ghent, Belgium